CLINICAL TRIAL: NCT03417271
Title: A Double-blind Randomized Crossover Comparison of Short Pulse Width Versus Conventional Pulse Width Deep Brain Stimulation (DBS) in Parkinson's Disease Patients With Previously Implanted DBS Systems- a Pilot Trial
Brief Title: Short Pulse Width DBS in Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 16/0772
Record Dates: First submitted 2018-01-17; First posted 2018-01-31 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Neither participants nor outcomes assessors will be aware whether the patient is receiving stimulation at 30us or 60us pulse widths.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 30us stimulation then 60us stimulation (Active Comparator): All patients will receive both types of stimulation in a randomised crossover design. This arm will receive 30us stimulation for 4 weeks then will be switched to 60us stimulation for 4 weeks.
  Interventions: Device: Deep brain stimulation
- 60us stimulation then 30us stimulation (Active Comparator): All patients will receive both types of stimulation in a randomised crossover design.This arm will receive 60us stimulation for 4 weeks then will be switched to 30us stimulation for 4 weeks.
  Interventions: Device: Deep brain stimulation

INTERVENTIONS:
Device: Deep brain stimulation — The different stimulation pulse widths are made possible by the use of a Medtronic XBP flashcard used with the conventional Medtronic 8840 programmer.

SUMMARY:
The aim of this investigation is to explore the effect of reducing conventional pulse width of stimulation on known adverse effects of Subthalamic nucleus Deep Brain Stimulation (STN DBS) treatment such as; slurring of speech, gait impairment, and unsteadiness. This investigation is designed such that each of 16 patients (who have all had chronically implanted DBS systems), will be assessed using conventional (DBS-60µs) and short (DBS-30µs) pulse width DBS, in a randomised order.

DETAILED DESCRIPTION:
Conventional DBS most commonly uses 60µs pulse width stimulation. Higher pulse widths are less well tolerated by patients as a result of adverse effects. The ability to use short pulse width (30µs) DBS in chronically implanted STN-DBS patients has been made possible as a result of the provision of a novel software flashcard (8870 XBP application card) developed by Medtronic, compatible with the routine Medtronic N'Vision 8870 Clinician Programmer. The Medtronic 8870-XBP flashcard will enable shorter pulse width (30µs) to be used with previously implanted conventional Medtronic DBS hardware, however this is not licensed at present.

The aim of this clinical investigation is to confirm the longevity of response and the clinical relevance of DBS-30µs versus DBS-60µs in DBS patients using "optimized" stimulation amplitudes for each pulse-width. This project will be conducted in patients with Parkinson's disease who have had long term bilateral sub thalamic nucleus Deep Brain Stimulation implants. As such, they will be regular attenders at the Unit of Functional Neurosurgery, National Hospital for Neurology & Neurosurgery, and will have had frequent previous attempts at adjusting their DBS parameters including overnight stays, and off- medication assessments to optimize motor function and minimize adverse effects. They will be familiar with all procedures to be used in this study. They will be aware that the objective of the study is to identify whether additional improvements in dysarthric speech can be achieved by the use of a short pulse width setting and therefore will be highly motivated to participate.

This investigation is designed such that each patient will be assessed under the DBS-30µs and DBS-60µs pulse width condition, in a randomised order. The patients and rating clinicians will be blinded to randomisation order. An unblinded clinician will be responsible for programming the stimulation. The use of a crossover design allows each patient to essentially act as their own control subject, and will maximise the ability to judge using paired statistical tests whether there is a consistent advantage in speech intelligibility using the shorter pulse width (DBS-30µs).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease - PD is a clinical diagnosis and is based on the opinion of the PI on site after review of the clinical history, examination findings and response to PD medication. The Queen Square brain bank criteria MAY be used to help assist in the diagnosis although this need not be a formal inclusion criteria, and the relevance of a positive family history of PD, or a confirmed genetic basis for an individual's symptoms will be evaluated in the context of other clinical features in determining diagnosis and eligibility.
* Male or Female.
* Treatment with subthalamic deep brain stimulation using Medtronic Activa PC hardware for at least 12 months.
* Experiencing stimulation-induced slurring of speech defined as scoring 50-80% speech intelligibility on the Assessment of Intelligibility of Speech scale.
* All patients will be ≥ 25 and ≤ 75 years of age.
* Documented informed consent to participate.

Exclusion Criteria:

* Patients unable to provide documented informed consent.
* Already actively participating in an investigation of a drug, device or surgical treatment for Parkinson's disease.
* Potential participants who lack the capacity to give informed consent.
* Any medical, psychiatric or other condition which in the investigator's opinion compromises the potential participant's ability to participate fully.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

PRIMARY OUTCOMES:
Speech Intelligibility test | 4 weeks
  Percentage of intelligible words spoken during formal speech assessment

SECONDARY OUTCOMES:
Movement Disorders Society Unified Parkinson's Disease Rating Scale | 4 weeks
  Validated movement scale for Parkinson's disease. Range 0-132. Higher scores indicate worse disability.
Dyskinesia Rating Scale | 4 weeks
  Validated dyskinesia rating scale. Range 0-104. Higher scores indicate worse disability.
Verbal Fluency | 4 weeks
  Number of words produced in 1 minute
Timed Motor tests | 4 weeks
  Walking and hand tapping

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Foltynie, MRCP PhD, Principal Investigator — UCL Institute of Neurology
Locations (1):
- UCL Institute of Neurology, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No